CLINICAL TRIAL: NCT01552863
Title: Open-Label, Single-Dose, Randomized, Crossover Study To Evaluate The Pharmacokinetics Of Oxycodone Following Oral Administration Of PF-00345439 Under Fed Conditions In Healthy Volunteers
Brief Title: A Study To Characterize The Pharmacokinetics Of Oxycodone In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4501018
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Pain
Keywords: pharmacokinetics; bioavailability; oxycodone.
MeSH Terms: conditions — Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment B (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment C (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment D (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment E (Experimental): Single dose of 5 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment F (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation A, single dose
  Arms: Treatment A
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation E, single dose
  Arms: Treatment B
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation F, single dose
  Arms: Treatment C
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation G, single dose
  Arms: Treatment D
Drug: Oxycodone — One capsule of 5 mg PF-00345439 Formulation TBD, single dose
  Arms: Treatment E
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation H, single dose
  Arms: Treatment F

SUMMARY:
This is an open-label (both the physician and healthy volunteer know which medication will be administered), single-dose, 6- dosing period study to characterize the pharmacokinetics of oxycodone (process by which oxycodone is absorbed, distributed, metabolized, and eliminated by the body). This study will consist of three parts that will take place over approximately 90 days. Part 1 of the study has 4 dosing periods, while Parts 2 and 3 have one dosing period each.

DETAILED DESCRIPTION:
This study will estimate the PK and relative BA of oxycodone following single oral 40-mg doses of 3 modified PF-00345439 Formulations E, F, and G compared with the reference PF-00345439 Formulation A under fed conditions in healthy volunteers in order to aid in selection of a final formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between 18 and 55 years of age (inclusive).

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* History of obstructive sleep apnea.
* Positive urine drug test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve from Time Zero to Extrapolated Infinite Time [AUC(0-inf)] | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, and 48 hours post-dose.
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, and 48 hours post-dose.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Oxycodone in Treatment E | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, and 48 hours post-dose.
Area Under the Curve from Time Zero to Extrapolated Infinite Time [AUC(0-inf)] of Oxycodone in Treatment E | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, and 48 hours post-dose.
Area Under the Curve from Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, and 48 hours post-dose.
Plasma Concentration 24 Hours Post-Dose (C24) | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, and 24 hours post-dose.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, and 48 hours post-dose.
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, and 48 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4501018&StudyName=A%20Study%20To%20Characterize%20The%20Pharmacokinetics%20Of%20Oxycodone%20In%20Healthy%20Volunteers